CLINICAL TRIAL: NCT04178408
Title: Registry to Study the Incidence, Phenotype, Risk Factors and Clinical Course of Inflammatory Bowel Disease in Zimbabwe
Brief Title: IBD Registry in a Sub-Saharan African Population
Status: Recruiting | Type: Observational
Sponsor: University of Zimbabwe (Other)
Collaborators: Swiss IBDnet (Unknown); University of Bern (Other)
Responsible Party: Sponsor
Other Study IDs: IBDZIM
Record Dates: First submitted 2019-11-25; First posted 2019-11-26 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Inflammatory Bowel Diseases; Ulcerative Colitis; Crohn Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — stool specimens, and germline DNA from peripheral blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Cases of inflammatory bowel disease
  Interventions: Other: No intervention
- Controls: Two controls per case. 1. Sibling or other second degree relative of similar age. 2. neighbourhood control matched for age
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The investigators intend to establish a prospective registry of patients diagnosed with inflammatory bowel disease at Parirenyatwa hospital in Harare, Zimbabwe. The study will periodically collect data on disease phenotype, disease course, and clinical management, and will biobank stool specimens and germline DNA. One relative, and an individual from the same neighbourhood will be also be recruited for a nested case-control study into risk factors of inflammatory bowel disease in this population.

DETAILED DESCRIPTION:
A prospective observational registry with a nested case-control study will be established at a gastrointestinal outpatient's clinic at a tertiary care hospital in Harare, Zimbabwe. The registry will recruit confirmed cases of inflammatory bowel disease from the clinic, other hospitals within and outside Harare, and from private practitioners. Two controls, a sibling or cousin, and an individual living in the same neighbourhood will also be recruited for each case. Demographic and clinical data will be obtained for all cases at baseline, after 6 months and annually thereafter. A questionnaire adapted from the International Organisation of IBD for risk factors of inflammatory bowel disease, and a food frequency questionnaire will be administered to all participants. Stool specimens, and germline DNA from peripheral blood will be biobanked in the Department of Medicine at the University of Zimbabwe. Preliminary data analysis will be carried out after at least 100 patients have been recruited. Descriptive statistics will be used to summarise data on demographic and phenotypic characteristics of inflammatory bowel disease, and incidence will be estimated for Harare. Risk factors for inflammatory bowel disease will be analysed using conditional logistic regression.

ELIGIBILITY:
Inclusion Criteria:

* Cases

  1. Any patient with confirmed inflammatory bowel disease
  2. Onset of disease ≥3 months ago.
* Controls

  1. Age ≥ 18 years (NB - cases younger than 18 will be excluded from case-control analysis
  2. One sibling or cousin (2nd degree) and one neighbourhood control.

Exclusion Criteria:

* Cases

  1. None
* Controls

  1. Suspected inflammatory bowel disease
  2. Unexplained gastrointestinal symptoms including diarrhoea, vomiting, chronic abdominal pain, weight loss, rectal bleeding, and recent change in bowel habit.
  3. Previous unexplained gastrointestinal surgery

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Cases of inflammatory bowel disease and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-01-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Demographic and phenotypic features of inflammatory bowel disease | one year
  Data on demographic (age, gender, ethnicity) and phenotypic (Crohn's disease versus ulcerative colitis, location, severity, extra-intestinal manifestations etc) will be collected using a standardised case report report forms

SECONDARY OUTCOMES:
Risk factors of inflammatory bowel disease in Zimbabwe | Two years
  Odds ratios of risk factors such as exposure to antibiotics, smoking, markers of hygiene such as sanitary conditions, etc) collected using the using the International Organisation for the Study of Inflammatory bowel disease (IOBD) risk factor questionnaire will be calculated.
Dietary risk factors of inflammatory bowel disease in Zimbabwe | Two years
  Odds ratios for dietary patterns derived from a validated semi-quantitative food frequency questionnaire administered to cases and controls will be calculated.
Incidence and prevalence of inflammatory bowel disease in Zimbabwe | Three years
  The incidence and prevalence will be estimated using the annual number of new cases, and the total number of cases in Harare respectively and the total population of the city as the denominator.

CONTACTS AND LOCATIONS:
Overall Officials: Leolin Katsidzira, MD, Principal Investigator — University of Zimbabwe
Locations (1):
- Parirenyatwa Hospital, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Katsidzira L, Mudombi WF, Makunike-Mutasa R, Yilmaz B, Blank A, Rogler G, Macpherson A, Vavricka S, Gangaidzo I, Misselwitz B. Inflammatory bowel disease in sub-Saharan Africa: a protocol of a prospective registry with a nested case-control study. BMJ Open. 2020 Dec 22;10(12):e039456. doi: 10.1136/bmjopen-2020-039456. PMID 33371021